CLINICAL TRIAL: NCT01258608
Title: A Randomized, Multi-Center, Blinded, Placebo-Controlled Study Of Mapatumumab ([HGS1012], A Fully Monoclonal Antibody To TRAIL-R1) In Combination With Sorafenib As A First-Line Therapy In Subjects With Advanced Hepatocellular Carcinoma
Brief Title: Study of Mapatumumab in Combination With Sorafenib in Subjects With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200149; HGS1012-C1103 (Other: Human Genome Sciences Inc.)
Record Dates: First submitted 2010-12-07; First posted 2010-12-13 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: advanced hepatocellular carcinoma; Mapatumumab; HGS1012; sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — mapatumumab; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib plus mapatumumab (Experimental): Mapatumumab 30 milligrams (mg)/kilogram (kg) intravenously on Day 1 of each cycle (i.e. every 21 days) plus sorafenib 400 mg orally twice daily continuously in each cycle until radiologic disease progression or unacceptable toxicity
  Interventions: Drug: Mapatumumab; Drug: Sorafenib
- Sorafenib plus Placebo (Placebo Comparator): Placebo intravenously on Day 1 of each cycle (i.e. every 21 days) plus sorafenib 400 mg orally twice daily continuously in each cycle until radiologic disease progression or unacceptable toxicity
  Interventions: Drug: Placebo; Drug: Sorafenib

INTERVENTIONS:
Drug: Mapatumumab — Mapatumumab will be supplied as a lyophilized formulation in 10 mL vials containing 100 mg mapatumumab for intravenous infusion at the dose of 30 mg/kg.
  Arms: Sorafenib plus mapatumumab
Drug: Placebo — Normal saline solution for intravenous infusion will be administered as placebo for mapatumumab
  Arms: Sorafenib plus Placebo
Drug: Sorafenib — Sorafenib will be supplied as tablets, each containing 274 mg sorafenib tosylate, equivalent to 200 mg of sorafenib, to be administered 400 mg (2 x 200 mg tablets) orally twice daily.

SUMMARY:
Mapatumumab is a fully human, agonist monoclonal antibody that activates the cell death pathway in tumor cells by specifically binding to TRAIL-R1 with high affinity. Sorafenib, a multikinase inhibitor, is the standard of care for treatment of patients with advanced hepatocellular carcinoma (HCC). The mechanisms of sorafenib and mapatumumab action suggest that these agents could interact synergistically. This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of mapatumumab in combination with sorafenib in subjects with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh Class A.
* Barcelona Clinic Liver Cancer (BCLC) advanced stage (C) hepatocellular carcinoma, or BCLC intermediate stage (B) hepatocellular carcinoma if treatment with transarterial chemoembolization is not considered appropriate
* Measurable disease demonstrating intratumoral arterial enhancement by contrast enhanced computerized tomography (CT), with use of multislice scanners, or contrast enhanced dynamic magnetic resonance imaging (MRI), with at least 1 tumor lesion that meets the following criteria: located in the liver; can be accurately measured in at least 1 dimension; well delineated area of viable, hypervascular (contrast enhancement in the arterial phase) tumor that is >2 centimeter (cm) in the axial plane; suitable for repeat measurement; OR not previously treated with locoregional or systemic treatment unless the lesion shows a well-delineated area of viable (contrast enhancement in the arterial phase) tumor that is >2 cm in the axial plane. (If the lesion is poorly demarcated or exhibits atypical enhancement as a result of the previous intervention, then it cannot be selected as a target lesion)
* Radiologic eligibility (measurable disease) must be must be confirmed by the BICR prior to randomization.
* Adequate bone marrow, renal and liver function as defined in the protocol.
* Performance status of 0, 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) Scale
* Age 18 years or older
* Have the ability to understand the requirements of the study, provide written informed consent (including consent for the use and disclosure of research-related health information), and comply with the study and follow-up procedures.

Exclusion Criteria:

* Any co-morbid condition that in the judgment of the investigator renders the subject at high risk of treatment complications or reduces the possibility of assessing clinical effect.
* Received prior investigational or non-investigational cytotoxic chemotherapy, hormonal therapy, biological therapy (including but not limited to monoclonal antibodies, small molecules or other immunotherapy) to treat hepatocellular carcinoma.
* History of organ allograft.
* Previously received mapatumumab or sorafenib.
* Underwent resection, radiofrequency ablation, radiation or chemoembolization within 4 weeks before enrollment or not recovered from such treatments.
* Need for concomitant anticancer therapy (surgery, radiation therapy, chemotherapy, immunotherapy, radiofrequency ablation) or other investigational agents during the study treatment period.
* Major surgery (i.e., the opening of a major body cavity, requiring the use of general anesthesia) within 4 weeks before enrollment; minor surgery (except for insertion of vascular access device) within 2 weeks before enrollment; or not yet recovered from the effects of the surgery.
* Systemic steroids within 1 week before enrollment except steroids used as part of an antiemetic regimen or maintenance-dose steroids for non-cancerous disease.
* Hepatic encephalopathy, per the investigator's evaluation.
* History of clinically significant gastrointestinal bleeding requiring procedural intervention (e.g., variceal banding, transjugular intrahepatic portosystemic shunt procedure, arterial embolization, topical coagulation therapy) within 4 weeks before enrollment.
* Gastrointestinal disease resulting in an inability to take oral medication or a requirement for intravenous hyperalimentation.
* History of any infection requiring hospitalization or intravenous antibiotics within 2 weeks before enrollment.
* Known brain or spinal cord metastases unless adequately treated (surgery or radiotherapy) with no evidence of progression and neurologically stable off anticonvulsants and steroids.
* Known human immunodeficiency virus infection.
* Unstable angina, myocardial infarction, cerebrovascular accident, >= Class II congestive heart failure according to the New York Heart Association Classification for Congestive Heart Failure within 6 months before enrollment.
* Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
* Uncontrolled hypertension (systolic blood pressure >150 millimeters of mercury [mmHg] or diastolic pressure >90 mmHg despite optimal medical management).
* Using and unable to discontinue use of concomitant strong CYP3A4 inducers (e.g., including but not limited to St. John's Wort, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, phenobarbital)
* Pregnant female or nursing mother. All females with an intact uterus (unless amenorrheic for the 24 months before enrollment) must have a negative serum pregnancy test at screening. All non-sterile or non-postmenopausal females must practice a medically accepted method of contraception over the course of the study and for 60 days after the last dose of study agent.
* Males who do not agree to use effective contraception during the study and for a period of 60 days following the final dose of study agent.
* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s) or subject is receiving other investigational agents.
* Acute or chronic severe renal insufficiency (glomoerular filtration rate <30 milliliters [mL]/minute/1.73 square meters) or acute renal insufficiency of any severity due to the hepato-renal syndrome.
* Hepatitis B virus deoxyribonucleic acid (DNA) levels >2,000 international units/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-02-08 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (37):
- United States (8):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Hamburg
- Poland (5):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, San Juan, Puerto Rico
- Romania (4):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Iași
- Russia (8):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
  - GSK Investigational Site, Uzhhorod
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ciuleanu T, Bazin I, Lungulescu D, Miron L, Bondarenko I, Deptala A, Rodriguez-Torres M, Giantonio B, Fox NL, Wissel P, Egger J, Ding M, Kalyani RN, Humphreys R, Gribbin M, Sun W. A randomized, double-blind, placebo-controlled phase II study to assess the efficacy and safety of mapatumumab with sorafenib in patients with advanced hepatocellular carcinoma. Ann Oncol. 2016 Apr;27(4):680-7. doi: 10.1093/annonc/mdw004. Epub 2016 Jan 22. PMID 26802147
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 200149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200149 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2, multi-center, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of mapatumumab in combination with sorafenib in participants with advanced hepatocellular carcinoma.
Pre-assignment Details: A total of 217 participants were screened of which 116 were screen failures and 101 participants were randomized in a ratio of 1:1 to any one of the 2 treatment arms. The study was conducted at 29 centers in 6 countries.
Groups:
- Sorafenib+Placebo: Participants received sorafenib 400 milligrams (mg) orally twice daily continuously in each 21-day cycle. Placebo was administered via the intravenous route on Day 1 of each 21-day cycle. The treatments were administered until radiologic disease progression or unacceptable toxicity
- Sorafenib+Mapatumumab 30 mg/kg: Participants received sorafenib 400 mg orally twice daily continuously in each 21-day cycle. Mapatumumab 30 milligrams per kilogram (mg/kg) was administered via the intravenous route on Day 1 of each 21-day cycle. The treatments were administered until radiologic disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Started | 51 | 50
Completed (Completed placebo/mapatumumab treatment defined as treated until radiologic disease progression) | 30 | 31
Not Completed | 21 | 19
Not completed — Metastatic Hepatocellular Carcinoma | 1 | 0
Not completed — Clinical progression | 1 | 0
Not completed — Sponsor decision | 0 | 1
Not completed — Physician Decision | 6 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of compliance | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 6 | 10
Not completed — Withdrawal by Subject | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (13.36) | 60.0 (11.93) | 60.4 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 24 | 36
  Male | 39 | 26 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian - European Heritage | 48 | 48 | 96
  Asian-East Asian Heritage | 1 | 0 | 1
  Black or African American | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression-Blinded Independent Central Review (BICR) Assessment
Description: Time to progression is defined as the time from randomization to radiologic disease progression based on blinded independent review (BICR) of imaging scans using modified Response Evaluation Criteria in Solid Tumors assessment (mRECIST) for hepatocellular carcinoma. The primary analysis was performed using Kaplan Meier methods. The median time to progression is reported with one-sided 90% confidence interval. Analysis was performed on the modified Intent to Treat (mITT) Population which comprised of all randomized participants who received at least part of 1 dose of study agent (mapatumumab/placebo and/or sorafenib) with participants analyzed according to the groups to which they were randomized. NA indicates upper limit was not measurable as one-sided confidence interval is presented.
Time Frame: Randomization to maximum of 24.1 months
Population: mITT Population. Only those participants who had their BICR scans read were included in the analysis.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 48 | 45
Months | 5.6 [4.3 to NA] — Upper limit was not measurable as one-sided confidence interval is presented | 4.1 [2.8 to NA] — Upper limit was not measurable as one-sided confidence interval is presented.
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.7382, Stratified log-rank test — P-value for comparison of treatment groups obtained from stratified log-rank test-stratified by Barcelona Clinic Liver Cancer and Eastern Cooperative Oncology Group (ECOG) performance status; Hazard Ratio (HR) = 1.192, 90% CI 1-sided [upper limit 1.737] — Hazard ratio comparing mapatumumab to placebo obtained from Cox proportional hazards model with covariate adjustment for Barcelona Clinic Liver Cancer and ECOG performance status

2. Secondary Outcome: Time to Progression-Investigator Assessment
Description: Time to progression is defined as the time from randomization to radiologic disease progression. The primary analysis was performed using Kaplan Meier methods based on application of mRECIST for hepatocellular carcinoma to investigator assessments. The median time to progression is reported with one-sided 90% confidence interval. NA indicates upper limit was not measurable as one-sided confidence interval is presented.
Time Frame: Randomization to maximum of 52.9 months
Population: mITT Population
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Months | 8.3 [5.4 to NA] — Upper limit was not measurable as one-sided confidence interval is presented. | 6.4 [5.4 to NA] — Upper limit was not measurable as one-sided confidence interval is presented.
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.3156, Stratified log-rank test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.922, 90% CI 1-sided [upper limit 1.288] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Median Overall Survival
Description: Overall survival is defined as time from randomization to death from any cause. The analysis was performed using Kaplan Meier methods. The median overall survival is reported with one-sided 90% confidence interval. NA indicates upper limit was not measurable as one-sided confidence interval is presented.
Time Frame: Randomization to maximum of 52.9 months
Population: mITT Population
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Months | 10.1 [8.9 to NA] — Upper limit was not measurable as one-sided confidence interval is presented. | 10.0 [7.3 to NA] — Upper limit was not measurable as one-sided confidence interval is presented.
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.6121, Stratified log-rank test — P-value for comparison of treatment groups obtained from stratified log-rank test-stratified by Barcelona Clinic Liver Cancer and ECOG performance status; Hazard Ratio (HR) = 1.007, 90% CI 1-sided [upper limit 1.346] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Progression Free Survival-BICR Assessment
Description: Progression free survival is defined as time from randomization to radiologic disease progression or death from any cause. The analysis was performed using Kaplan Meier methods using BICR assessment of imaging scans. The median progression free survival is reported with one-sided 90% confidence interval. NA indicates upper limit was not measurable as one-sided confidence interval is presented.
Time Frame: Randomization to maximum of 24.1 months
Population: mITT Population. Only those participants who had their BICR scans read were included in the analysis.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 48 | 45
Months | 4.3 [3.1 to NA] — Upper limit was not measurable as one-sided confidence interval is presented. | 3.2 [2.7 to NA] — Upper limit was not measurable as one-sided confidence interval is presented.
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.6925, Stratified log-rank test — P-value for comparison of treatment groups obtained from stratified log-rank test - stratified by Barcelona Clinic Liver Cancer and ECOG performance status; Hazard Ratio (HR) = 1.066, 90% CI 1-sided [upper limit 1.430] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Progression Free Survival-Investigator Assessment
Description: Progression free survival is defined as time from randomization to radiologic disease progression or death from any cause. The analysis was performed using Kaplan Meier methods based on application of mRECIST for hepatocellular carcinoma to investigator assessments. The median progression free survival is reported with one-sided 90% confidence interval. NA indicates upper limit was not measurable as one-sided confidence interval is presented.
Time Frame: Randomization to maximum of 52.9 months
Population: mITT Population
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Months | 5.4 [3.6 to NA] — Upper limit was not measurable as one-sided confidence interval is presented. | 4.0 [3.4 to NA] — Upper limit was not measurable as one-sided confidence interval is presented.
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.3088, Stratified log-rank test — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.909, 90% CI 1-sided [upper limit 1.191] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percentage of Participants With Objective Response-BICR Assessment
Description: Objective response rate is defined as the percentage of participants with complete response+partial response according to mRECIST criteria for hepatocellular carcinoma using BICR assessment of imaging scans. The percentage of participants with objective response is reported along with 95% confidence interval.
Time Frame: Randomization to maximum of 24.1 months
Population: mITT Population. Only those participants who had their BICR scans read and having available assessment for best response were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 40 | 39
Percentage of participants | 12.5 [4.2 to 26.8] | 17.9 [7.5 to 33.5]
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.5458, Fisher Exact — Nominal P-value for comparison of treatment groups obtained from Fisher's exact test; Response rate difference = 5.4, 95% CI 2-sided [-16.8 to 26.6]

7. Secondary Outcome: Percentage of Participants With Objective Response-Investigator Assessment
Description: Objective response rate is defined as the percentage of participants with complete response+partial response according to mRECIST criteria for hepatocellular carcinoma to investigator assessments. The percentage of participants with objective response is reported along with 95% confidence interval.
Time Frame: Randomization to maximum of 52.9 months
Population: mITT Population. Only those participants with available assessment for best response were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 48
Percentage of participants | 7.8 [2.2 to 18.9] | 14.6 [6.1 to 27.8]
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.3479, Fisher Exact — Nominal P-value for comparison of treatment groups obtained from Fisher's exact test; Response rate difference = 6.7, 95% CI 2-sided [-13.4 to 26.2]

8. Secondary Outcome: Percentage of Participants With Disease Control-BICR Assessment
Description: Disease control rate is the percentage of participants with complete response+partial response+stable disease according to mRECIST criteria for hepatocellular carcinoma. The end point was based on BICR assessment of imaging scans. The percentage of participants with disease control is presented along with 95% confidence interval.
Time Frame: Randomization to maximum of 24.1 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 40 | 39
Percentage of participants | 92.5 [79.6 to 98.4] | 71.8 [55.1 to 85.0]
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.0198, Fisher Exact — Nominal P-value for comparison of treatment groups obtained from Fisher's exact test; Disease control rate difference = -20.7, 95% CI 2-sided [-40.8 to 1.8]

9. Secondary Outcome: Percentage of Participants With Disease Control-Investigator Assessment
Description: Disease control rate is the percentage of participants with complete response+partial response+stable disease according to mRECIST criteria for hepatocellular carcinoma to investigator assessments. The percentage of participants with disease control is presented along with 95% confidence interval.
Time Frame: Randomization to maximum of 52.9 months
Population: mITT Population. Only those participants with available assessment for best response were analyzed
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 48
Percentage of participants | 74.5 [60.4 to 85.7] | 68.8 [53.7 to 81.3]
Statistical Analysis 1: Comparison: Sorafenib+Placebo vs Sorafenib+Mapatumumab 30 mg/kg; Test type: Other; p = 0.6558, Fisher Exact — Nominal P-value for comparison of treatment groups obtained from Fisher's exact test; Disease control rate difference = -5.8, 95% CI 2-sided [-25.4 to 13.8]

10. Secondary Outcome: Time to Response-BICR Assessment
Description: Time to response is defined as time from randomization to first partial response or complete response in responders only. Complete Response (CR): Disappearance of intratumoral arterial enhancement in all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions
Time Frame: Randomization to maximum of 24.1 months
Population: mITT Population. Only responders were included in the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 5 | 7
Days | 44 [41 to 85] | 48 [41 to 188]

11. Secondary Outcome: Duration of Response-BICR Assessment
Description: Duration of response is defined as time from first PR or CR to radiologic disease progression; in responders only. CR: Disappearance of intratumoral arterial enhancement in all target lesions. PR: At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the Baseline sum of the diameters of target lesions. Progressive disease (PD): An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started.
Time Frame: Randomization to maximum of 24.1 months
Population: mITT Population. Only responders were included in the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 5 | 7
Days | 123 [55 to 325] | 127 [42 to 372]

12. Secondary Outcome: Number of Participants With Treatment-emergent Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any unfavorable or unintended sign, symptom, or disease that is temporally associated with the use of a study agent but is not necessarily caused by the study agent. An SAE is an adverse event resulting in any of the following outcomes: death, life-threatening, inpatient hospitalization, prolongation of an existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect or other medically important events that may jeopardize the participant or may require intervention to prevent one of the other outcomes mentioned before. A treatment-emergent AE is an AE that emerged during treatment, having been absent pre-treatment, or worsened relative to the pre-treatment state. As-Treated Population comprised of participants who received at least part of 1 dose of study agent analyzed according to the treatment that they actually received.
Time Frame: Start of study treatment to maximum of 52.9 months
Population: As-Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Participants
  Non-serious AEs | 47 | 49
  SAEs | 27 | 21

13. Secondary Outcome: Number of Participants With Severe AEs
Description: An AE is any unfavorable or unintended sign, symptom, or disease that is temporally associated with the use of a study agent but is not necessarily caused by the study agent. Severity of AEs were graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0. Grade 1 represents mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 represents moderate; minimal, local or non-invasive intervention indicated. Grade 3 represents severe or medically significant but not immediately life -threatening; hospitalization or prolongation of hospitalization indicated; disabling. Grade 4 represents life -threatening consequences; urgent intervention indicated. Grade 5 represents death related to AE. Severe AE is defined as AEs classified by investigator as severe (causing inability to carry out usual activities), life threatening or fatal using NCI-CTCAE Version 4.0 grading.
Time Frame: Start of study treatment to maximum of 52.9 months
Population: As-Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Participants | 42 | 38

14. Secondary Outcome: Number of Participants With Worst Toxicity Grade-chemistry Parameters
Description: Blood samples were collected for the evaluation of following chemistry parameters: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), amylase, bilirubin, gamma glutamyl transferase (GGT), calcium, potassium, magnesium, albumin, sodium and creatinine. Laboratory toxicities were graded based on the NCI-CTCAE version 4.0. Grade 1 represents mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 represents moderate; minimal, local or non-invasive intervention indicated. Grade 3 represents severe or medically significant but not immediately life -threatening; hospitalization or prolongation of hospitalization indicated; disabling. Grade 4 represents life -threatening consequences; urgent intervention indicated. Number of participants with worst toxicity grades for any abnormalities observed in any chemistry parameters during the study is presented.
Time Frame: Enrolment to maximum of 52.9 months
Population: As-Treated Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Participants
  ALT increased; Grade 0, n=51, 50 | 6 | 4
  ALT increased; Grade 1, n=51, 50 | 30 | 28
  ALT increased; Grade 2, n=51, 50 | 8 | 9
  ALT increased; Grade 3, n=51, 50 | 7 | 9
  ALT increased; Grade 4, n=51, 50 | 0 | 0
  AST increased; Grade 0, n=51, 50 | 1 | 1
  AST increased; Grade 1, n=51, 50 | 23 | 20
  AST increased; Grade 2, n=51, 50 | 10 | 9
  AST increased; Grade 3, n=51, 50 | 16 | 20
  AST increased; Grade 4, n=51, 50 | 1 | 0
  ALP increased; Grade 0, n=51, 50 | 4 | 8
  ALP increased; Grade 1, n=51, 50 | 31 | 26
  ALP increased; Grade 2, n=51, 50 | 11 | 11
  ALP increased; Grade 3, n=51, 50 | 5 | 5
  ALP increased; Grade 4, n=51, 50 | 0 | 0
  Amylase increased; Grade 0, n=51, 50 | 30 | 22
  Amylase increased; Grade 1, n=51, 50 | 9 | 17
  Amylase increased; Grade 2, n=51, 50 | 5 | 8
  Amylase increased; Grade 3, n=51, 50 | 6 | 3
  Amylase increased; Grade 4, n=51, 50 | 1 | 0
  Bilirubin increased; Grade 0, n=51, 50 | 12 | 9
  Bilirubin increased; Grade 1, n=51, 50 | 15 | 10
  Bilirubin increased; Grade 2, n=51, 50 | 17 | 16
  Bilirubin increased; Grade 3, n=51, 50 | 7 | 13
  Bilirubin increased; Grade 4, n=51, 50 | 0 | 2
  GGT increased; Grade 0, n=51, 50 | 1 | 2
  GGT increased; Grade 1, n=51, 50 | 10 | 13
  GGT increased; Grade 2, n=51, 50 | 14 | 15
  GGT increased; Grade 3, n=51, 50 | 23 | 18
  GGT increased; Grade 4, n=51, 50 | 3 | 2
  Hypercalcemia; Grade 0, n=49, 47: number analyzed (Participants) | 49 | 47
  Hypercalcemia; Grade 0, n=49, 47 | 37 | 37
  Hypercalcemia; Grade 1, n=49, 47: number analyzed (Participants) | 49 | 47
  Hypercalcemia; Grade 1, n=49, 47 | 11 | 9
  Hypercalcemia; Grade 2, n=49, 47: number analyzed (Participants) | 49 | 47
  Hypercalcemia; Grade 2, n=49, 47 | 1 | 0
  Hypercalcemia; Grade 3, n=49, 47: number analyzed (Participants) | 49 | 47
  Hypercalcemia; Grade 3, n=49, 47 | 0 | 0
  Hypercalcemia; Grade 4, n=49, 47: number analyzed (Participants) | 49 | 47
  Hypercalcemia; Grade 4, n=49, 47 | 0 | 1
  Hyperkalemia; Grade 0; n=51, 50 | 36 | 27
  Hyperkalemia; Grade 1; n=51, 50 | 2 | 3
  Hyperkalemia; Grade 2; n=51, 50 | 10 | 10
  Hyperkalemia; Grade 3; n=51, 50 | 0 | 7
  Hyperkalemia; Grade 4; n=51, 50 | 3 | 3
  Hypermagnesemia; Grade 0; n=51, 50 | 29 | 28
  Hypermagnesemia; Grade 1; n=51, 50 | 21 | 19
  Hypermagnesemia; Grade 2; n=51, 50 | 0 | 0
  Hypermagnesemia; Grade 3; n=51, 50 | 1 | 3
  Hypermagnesemia; Grade 4; n=51, 50 | 0 | 0
  Hypernatremia; Grade 0, n=51, 50 | 18 | 18
  Hypernatremia; Grade 1, n=51, 50 | 16 | 14
  Hypernatremia; Grade 2, n=51, 50 | 0 | 0
  Hypernatremia; Grade 3, n=51, 50 | 16 | 15
  Hypernatremia; Grade 4, n=51, 50 | 1 | 3
  Hypoalbuminemia; Grade 0, n=51, 50 | 22 | 26
  Hypoalbuminemia; Grade 1, n=51, 50 | 10 | 9
  Hypoalbuminemia; Grade 2, n=51, 50 | 18 | 14
  Hypoalbuminemia; Grade 3, n=51, 50 | 1 | 1
  Hypoalbuminemia; Grade 4, n=51, 50 | 0 | 0
  Hypocalcemia; Grade 0, n=50, 50: number analyzed (Participants) | 50 | 50
  Hypocalcemia; Grade 0, n=50, 50 | 16 | 15
  Hypocalcemia; Grade 1, n=50, 50: number analyzed (Participants) | 50 | 50
  Hypocalcemia; Grade 1, n=50, 50 | 8 | 14
  Hypocalcemia; Grade 2, n=50, 50: number analyzed (Participants) | 50 | 50
  Hypocalcemia; Grade 2, n=50, 50 | 18 | 19
  Hypocalcemia; Grade 3, n=50, 50: number analyzed (Participants) | 50 | 50
  Hypocalcemia; Grade 3, n=50, 50 | 6 | 2
  Hypocalcemia; Grade 4, n=50, 50: number analyzed (Participants) | 50 | 50
  Hypocalcemia; Grade 4, n=50, 50 | 2 | 0
  Hypokalemia; Grade 0, n=51, 50 | 37 | 41
  Hypokalemia; Grade 1, n=51, 50 | 11 | 8
  Hypokalemia; Grade 2, n=51, 50 | 0 | 0
  Hypokalemia; Grade 3, n=51, 50 | 1 | 1
  Hypokalemia; Grade 4, n=51, 50 | 2 | 0
  Hypomagnesemia; Grade 0, n=51, 50 | 30 | 35
  Hypomagnesemia; Grade 1, n=51, 50 | 19 | 13
  Hypomagnesemia; Grade 2, n=51, 50 | 2 | 1
  Hypomagnesemia; Grade 3, n=51, 50 | 0 | 0
  Hypomagnesemia; Grade 4, n=51, 50 | 0 | 1
  Hyponatremia; Grade 0, n=49, 47: number analyzed (Participants) | 49 | 47
  Hyponatremia; Grade 0, n=49, 47 | 40 | 32
  Hyponatremia; Grade 1, n=49, 47: number analyzed (Participants) | 49 | 47
  Hyponatremia; Grade 1, n=49, 47 | 5 | 10
  Hyponatremia; Grade 2, n=49, 47: number analyzed (Participants) | 49 | 47
  Hyponatremia; Grade 2, n=49, 47 | 2 | 3
  Hyponatremia; Grade 3, n=49, 47: number analyzed (Participants) | 49 | 47
  Hyponatremia; Grade 3, n=49, 47 | 2 | 2
  Hyponatremia; Grade 4, n=49, 47: number analyzed (Participants) | 49 | 47
  Hyponatremia; Grade 4, n=49, 47 | 0 | 0
  Lipase increased; Grade 0, n=51, 50 | 19 | 13
  Lipase increased; Grade 1, n=51, 50 | 5 | 6
  Lipase increased; Grade 2, n=51, 50 | 8 | 8
  Lipase increased; Grade 3, n=51, 50 | 16 | 17
  Lipase increased; Grade 4, n=51, 50 | 3 | 6
  Renal: Creatinine increased; Grade 0, n=51, 50 | 36 | 34
  Renal: Creatinine increased; Grade 1, n=51, 50 | 7 | 12
  Renal: Creatinine increased; Grade 2, n=51, 50 | 8 | 3
  Renal: Creatinine increased; Grade 3, n=51, 50 | 0 | 1
  Renal: Creatinine increased; Grade 4, n=51, 50 | 0 | 0

15. Secondary Outcome: Number of Participants With Worst Toxicity Grade-hematology Parameters
Description: Blood samples were collected for assessment of the following hematology parameters: activated partial thromboplastin time (APTT), hemoglobin, international normalized ratio (INR), lymphocytes, neutrophils, platelets and white blood cells (WBC). Laboratory toxicities were graded based on the NCI-CTCAE version 4.0. Grade 1 represents mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 represents moderate; minimal, local or non-invasive intervention indicated. Grade 3 represents severe or medically significant but not immediately life -threatening; hospitalization or prolongation of hospitalization indicated; disabling. Grade 4 represents life -threatening consequences; urgent intervention indicated. Number of participants with worst toxicity grades for any abnormalities observed in any hematology parameters during the study is presented.
Time Frame: Enrolment to maximum of 52.9 months
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Participants
  APTT prolonged; Grade 0, n=51, 50 | 24 | 22
  APTT prolonged; Grade 1, n=51, 50 | 19 | 24
  APTT prolonged; Grade 2, n=51, 50 | 6 | 2
  APTT prolonged; Grade 3, n=51, 50 | 2 | 2
  APTT prolonged; Grade 4, n=51, 50 | 0 | 0
  Anemia; Grade 0, n=51, 50 | 13 | 9
  Anemia; Grade 1, n=51, 50 | 23 | 22
  Anemia; Grade 2, n=51, 50 | 9 | 16
  Anemia; Grade 3, n=51, 50 | 6 | 3
  Anemia; Grade 4, n=51, 50 | 0 | 0
  Hemoglobin increased; Grade 0, n=46, 44: number analyzed (Participants) | 46 | 44
  Hemoglobin increased; Grade 0, n=46, 44 | 46 | 44
  Hemoglobin increased; Grade 1, n=46, 44: number analyzed (Participants) | 46 | 44
  Hemoglobin increased; Grade 1, n=46, 44 | 0 | 0
  Hemoglobin increased; Grade 2, n=46, 44: number analyzed (Participants) | 46 | 44
  Hemoglobin increased; Grade 2, n=46, 44 | 0 | 0
  Hemoglobin increased; Grade 3, n=46, 44: number analyzed (Participants) | 46 | 44
  Hemoglobin increased; Grade 3, n=46, 44 | 0 | 0
  Hemoglobin increased; Grade 4, n=46, 44: number analyzed (Participants) | 46 | 44
  Hemoglobin increased; Grade 4, n=46, 44 | 0 | 0
  INR increased; Grade 0, n=51, 50 | 2 | 3
  INR increased; Grade 1, n=51, 50 | 35 | 30
  INR increased; Grade 2, n=51, 50 | 12 | 14
  INR increased; Grade 3, n=51, 50 | 2 | 3
  INR increased; Grade 4, n=51, 50 | 0 | 0
  Lymphocytes decreased; Grade 0, n=51, 50 | 24 | 23
  Lymphocytes decreased; Grade 1, n=51, 50 | 3 | 0
  Lymphocytes decreased; Grade 2, n=51, 50 | 16 | 18
  Lymphocytes decreased; Grade 3, n=51, 50 | 8 | 8
  Lymphocytes decreased; Grade 4, n=51, 50 | 0 | 1
  Lymphocytes increased; Grade 0, n=51, 49: number analyzed (Participants) | 51 | 49
  Lymphocytes increased; Grade 0, n=51, 49 | 49 | 45
  Lymphocytes increased; Grade 1, n=51, 49: number analyzed (Participants) | 51 | 49
  Lymphocytes increased; Grade 1, n=51, 49 | 0 | 0
  Lymphocytes increased; Grade 2, n=51, 49: number analyzed (Participants) | 51 | 49
  Lymphocytes increased; Grade 2, n=51, 49 | 2 | 4
  Lymphocytes increased; Grade 3, n=51, 49: number analyzed (Participants) | 51 | 49
  Lymphocytes increased; Grade 3, n=51, 49 | 0 | 0
  Lymphocytes increased; Grade 4, n=51, 49: number analyzed (Participants) | 51 | 49
  Lymphocytes increased; Grade 4, n=51, 49 | 0 | 0
  Neutrophil count decreased; Grade 0, n=51, 50 | 39 | 37
  Neutrophil count decreased; Grade 1, n=51, 50 | 3 | 2
  Neutrophil count decreased; Grade 2, n=51, 50 | 8 | 7
  Neutrophil count decreased; Grade 3, n=51, 50 | 1 | 1
  Neutrophil count decreased; Grade 4, n=51, 50 | 0 | 3
  Platelets decreased; Grade 0, n=51, 50 | 21 | 21
  Platelets decreased; Grade 1, n=51, 50 | 12 | 16
  Platelets decreased; Grade 2, n=51, 50 | 10 | 6
  Platelets decreased; Grade 3, n=51, 50 | 7 | 5
  Platelets decreased; Grade 4, n=51, 50 | 1 | 2
  WBC decreased; Grade 0, n=51, 50 | 33 | 30
  WBC decreased; Grade 1, n=51, 50 | 10 | 12
  WBC decreased; Grade 2, n=51, 50 | 8 | 5
  WBC decreased; Grade 3, n=51, 50 | 0 | 3
  WBC decreased; Grade 4, n=51, 50 | 0 | 0

16. Secondary Outcome: Number of Participants With Anti-mapatumumab Antibodies
Description: Blood samples were collected for the assessment of serum antibodies. The presence of anti-mapatumumab antibodies was assessed using a validated electrochemiluminescent immunoassay. The assay incorporated a tiered testing approach which used screening and confirmation steps. The anti-drug antibody (ADA) confirmed positive participants were separated into transient or persistent antibody positives. Persistent positive refers to positive immunogenic response at 2 or more assessments or at the final assessment. Transient positive refers to positive immunogenic response at only 1 assessment and negative at the final assessment.
Time Frame: Randomization to maximum of 24.1 months
Population: As-Treated Population. Only participants with an available immunogenicity assay were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 49
Participants
  Transient positive | 6
  Persistent positive | 7
  Negative | 36

17. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were obtained on Day 1 of each cycle. Baseline is the last assessment prior to first dose. Change from Baseline is the value at indicated time point minus the value at Baseline. NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time point.
Time Frame: Baseline and Day 1 of Cycles 2 to 75 (each cycle of 21 days)
Population: As Treated Population. Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Millimeters of mercury (mmHg)
  SBP; Cycle 2 Day 1, n=46, 44: number analyzed (Participants) | 46 | 44
  SBP; Cycle 2 Day 1, n=46, 44 | 2.3 (14.13) | 2.2 (18.64)
  SBP; CYCLE 3 DAY 1, n=39, 35: number analyzed (Participants) | 39 | 35
  SBP; CYCLE 3 DAY 1, n=39, 35 | 6.0 (16.81) | 4.1 (13.66)
  SBP; CYCLE 4; DAY 1; n=33, 32: number analyzed (Participants) | 33 | 32
  SBP; CYCLE 4; DAY 1; n=33, 32 | 2.1 (15.57) | 5.3 (13.52)
  SBP; CYCLE 5 DAY 1; n=27, 26: number analyzed (Participants) | 27 | 26
  SBP; CYCLE 5 DAY 1; n=27, 26 | 1.7 (13.05) | 4.9 (16.42)
  SBP; CYCLE 6 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  SBP; CYCLE 6 DAY 1; n=24, 22 | 1.3 (12.14) | 5.1 (13.40)
  SBP; CYCLE 7 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  SBP; CYCLE 7 DAY 1; n=24, 22 | -0.8 (11.02) | 5.0 (12.78)
  SBP; CYCLE 8 DAY 1; n=22, 21: number analyzed (Participants) | 22 | 21
  SBP; CYCLE 8 DAY 1; n=22, 21 | -1.6 (11.48) | 5.2 (14.83)
  SBP; CYCLE 9 DAY 1; n=19, 16: number analyzed (Participants) | 19 | 16
  SBP; CYCLE 9 DAY 1; n=19, 16 | 1.2 (16.37) | 7.8 (13.98)
  SBP; CYCLE 10 DAY 1; n=18, 16: number analyzed (Participants) | 18 | 16
  SBP; CYCLE 10 DAY 1; n=18, 16 | 1.4 (16.57) | 4.5 (16.19)
  SBP; CYCLE 11 DAY 1; n=16, 15: number analyzed (Participants) | 16 | 15
  SBP; CYCLE 11 DAY 1; n=16, 15 | 2.4 (18.82) | 5.2 (18.32)
  SBP; CYCLE 12 DAY 1; n=15, 13: number analyzed (Participants) | 15 | 13
  SBP; CYCLE 12 DAY 1; n=15, 13 | 2.7 (12.34) | 5.2 (14.73)
  SBP; CYCLE 13 DAY 1; n=13, 12: number analyzed (Participants) | 13 | 12
  SBP; CYCLE 13 DAY 1; n=13, 12 | 2.3 (12.26) | 3.0 (14.91)
  SBP; CYCLE 14 DAY 1; n=12, 12: number analyzed (Participants) | 12 | 12
  SBP; CYCLE 14 DAY 1; n=12, 12 | -1.0 (10.13) | 4.0 (14.63)
  SBP; CYCLE 15 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  SBP; CYCLE 15 DAY 1; n=10, 9 | 1.4 (8.21) | 6.7 (21.05)
  SBP; CYCLE 16 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  SBP; CYCLE 16 DAY 1; n=10, 9 | 1.8 (5.79) | 7.9 (15.28)
  SBP; CYCLE 17 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  SBP; CYCLE 17 DAY 1; n=8, 8 | 1.3 (11.95) | 10.1 (17.70)
  SBP; CYCLE 18 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  SBP; CYCLE 18 DAY 1; n=8, 8 | -2.0 (9.26) | 9.5 (19.41)
  SBP; CYCLE 19 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  SBP; CYCLE 19 DAY 1; n=6, 8 | -4.8 (14.93) | 8.4 (20.68)
  SBP; CYCLE 20 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  SBP; CYCLE 20 DAY 1; n=6, 8 | 1.2 (9.13) | 5.8 (19.33)
  SBP; CYCLE 21 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  SBP; CYCLE 21 DAY 1; n=4, 8 | 2.5 (8.23) | 10.0 (21.23)
  SBP; CYCLE 22 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  SBP; CYCLE 22 DAY 1; n=4, 8 | 6.0 (10.55) | 5.5 (14.11)
  SBP; CYCLE 23 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  SBP; CYCLE 23 DAY 1; n=4, 8 | -1.0 (10.80) | 12.9 (20.15)
  SBP; CYCLE 24 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  SBP; CYCLE 24 DAY 1; n=4, 8 | -3.0 (6.38) | 5.6 (19.86)
  SBP; CYCLE 25 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  SBP; CYCLE 25 DAY 1; n=4, 8 | 1.3 (12.20) | 11.3 (20.08)
  SBP; CYCLE 26 DAY 1; n=4, 7: number analyzed (Participants) | 4 | 7
  SBP; CYCLE 26 DAY 1; n=4, 7 | 6.0 (11.89) | 9.3 (22.92)
  SBP; CYCLE 27 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  SBP; CYCLE 27 DAY 1; n=4, 5 | 3.3 (10.44) | 8.4 (18.04)
  SBP; CYCLE 28 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  SBP; CYCLE 28 DAY 1; n=4, 5 | 3.3 (7.41) | 5.2 (20.19)
  SBP; CYCLE 29 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  SBP; CYCLE 29 DAY 1; n=3, 4 | -0.7 (14.29) | 3.3 (24.27)
  SBP; CYCLE 30 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  SBP; CYCLE 30 DAY 1; n=3, 4 | 2.7 (6.43) | -2.3 (13.43)
  SBP; CYCLE 31 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  SBP; CYCLE 31 DAY 1; n=3, 4 | -3.0 (11.79) | 2.0 (23.15)
  SBP; CYCLE 32 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  SBP; CYCLE 32 DAY 1; n=3, 4 | 5.0 (4.58) | 3.3 (16.40)
  SBP; CYCLE 33 DAY 1; n=2, 4: number analyzed (Participants) | 2 | 4
  SBP; CYCLE 33 DAY 1; n=2, 4 | 0.0 (14.14) | -5.3 (19.96)
  SBP; CYCLE 34 DAY 1; n=1, 4: number analyzed (Participants) | 1 | 4
  SBP; CYCLE 34 DAY 1; n=1, 4 | 13.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point. | -5.3 (10.66)
  SBP; CYCLE 35 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  SBP; CYCLE 35 DAY 1; n=0, 4 |  | -5.0 (15.81)
  SBP; CYCLE 36 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  SBP; CYCLE 36 DAY 1; n=0, 4 |  | -1.5 (13.00)
  SBP; CYCLE 37 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  SBP; CYCLE 37 DAY 1; n=0, 3 |  | -6.0 (23.52)
  SBP; CYCLE 38 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  SBP; CYCLE 38 DAY 1; n=0, 3 |  | -1.3 (18.04)
  SBP; CYCLE 39 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  SBP; CYCLE 39 DAY 1; n=0, 3 |  | -4.3 (21.01)
  SBP; CYCLE 40 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 40 DAY 1; n=0, 2 |  | -12.5 (10.61)
  SBP; CYCLE 41 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 41 DAY 1; n=0, 2 |  | -15.0 (21.21)
  SBP; CYCLE 42 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 42 DAY 1; n=0, 2 |  | -7.5 (17.68)
  SBP; CYCLE 43 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 43 DAY 1; n=0, 2 |  | -17.5 (17.68)
  SBP; CYCLE 44 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 44 DAY 1; n=0, 2 |  | -10.0 (14.14)
  SBP; CYCLE 45 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 45 DAY 1; n=0, 2 |  | -17.5 (17.68)
  SBP; CYCLE 46 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 46 DAY 1; n=0, 2 |  | -5.0 (21.21)
  SBP; CYCLE 47 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 47 DAY 1; n=0, 2 |  | -17.5 (17.68)
  SBP; CYCLE 48 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 48 DAY 1; n=0, 2 |  | -5.0 (21.21)
  SBP; CYCLE 49 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 49 DAY 1; n=0, 2 |  | -17.5 (17.68)
  SBP; CYCLE 50 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 50 DAY 1; n=0, 2 |  | -15.0 (21.21)
  SBP; CYCLE 51 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 51 DAY 1; n=0, 2 |  | -10.0 (21.21)
  SBP; CYCLE 52 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 52 DAY 1; n=0, 2 |  | -17.5 (17.68)
  SBP; CYCLE 53 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 53 DAY 1; n=0, 2 |  | -20.0 (14.14)
  SBP; CYCLE 54 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  SBP; CYCLE 54 DAY 1; n=0, 2 |  | -10.0 (14.14)
  SBP; CYCLE 55 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 55 DAY 1; n=0, 1 |  | -30.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 56 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 56 DAY 1; n=0, 1 |  | -30.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 57 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 57 DAY 1; n=0, 1 |  | -30.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 58 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 58 DAY 1; n=0, 1 |  | -25.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 59 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 59 DAY 1; n=0, 1 |  | -20.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 60 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 60 DAY 1; n=0, 1 |  | -30.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 61 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 61 DAY 1; n=0, 1 |  | -25.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 62 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 62 DAY 1; n=0, 1 |  | -23.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 63 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 63 DAY 1; n=0, 1 |  | -28.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 64 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 64 DAY 1; n=0, 1 |  | -25.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 65 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 65 DAY 1; n=0, 1 |  | -26.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 66 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 66 DAY 1; n=0, 1 |  | -32.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 67 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 67 DAY 1; n=0, 1 |  | -33.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 68 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 68 DAY 1; n=0, 1 |  | -32.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 69 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 69 DAY 1; n=0, 1 |  | -31.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 70 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 70 DAY 1; n=0, 1 |  | -25.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 71 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 71 DAY 1; n=0, 1 |  | -28.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 72 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 72 DAY 1; n=0, 1 |  | -30.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 73 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 73 DAY 1; n=0, 1 |  | -27.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 74 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 74 DAY 1; n=0, 1 |  | -30.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  SBP; CYCLE 75 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  SBP; CYCLE 75 DAY 1; n=0, 1 |  | -28.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; Cycle 2 Day 1, n=46, 44: number analyzed (Participants) | 46 | 44
  DBP; Cycle 2 Day 1, n=46, 44 | -0.6 (8.51) | 0.7 (9.82)
  DBP; CYCLE 3 DAY 1, n=39, 35: number analyzed (Participants) | 39 | 35
  DBP; CYCLE 3 DAY 1, n=39, 35 | 2.1 (7.20) | 1.4 (8.90)
  DBP; CYCLE 4; DAY 1; n=33, 32: number analyzed (Participants) | 33 | 32
  DBP; CYCLE 4; DAY 1; n=33, 32 | 1.8 (10.52) | 2.4 (8.22)
  DBP; CYCLE 5 DAY 1; n=27, 26: number analyzed (Participants) | 27 | 26
  DBP; CYCLE 5 DAY 1; n=27, 26 | 0.9 (10.00) | 3.0 (15.49)
  DBP; CYCLE 6 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  DBP; CYCLE 6 DAY 1; n=24, 22 | 3.5 (8.32) | 1.2 (10.21)
  DBP; CYCLE 7 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  DBP; CYCLE 7 DAY 1; n=24, 22 | 0.5 (8.57) | 2.0 (7.42)
  DBP; CYCLE 8 DAY 1; n=22, 21: number analyzed (Participants) | 22 | 21
  DBP; CYCLE 8 DAY 1; n=22, 21 | 0.5 (7.37) | 2.3 (8.27)
  DBP; CYCLE 9 DAY 1; n=19, 16: number analyzed (Participants) | 19 | 16
  DBP; CYCLE 9 DAY 1; n=19, 16 | 2.7 (8.67) | 4.1 (9.15)
  DBP; CYCLE 10 DAY 1; n=18, 16: number analyzed (Participants) | 18 | 16
  DBP; CYCLE 10 DAY 1; n=18, 16 | 2.7 (9.81) | 2.4 (7.50)
  DBP; CYCLE 11 DAY 1; n=16, 15: number analyzed (Participants) | 16 | 15
  DBP; CYCLE 11 DAY 1; n=16, 15 | -0.1 (10.25) | 0.9 (9.49)
  DBP; CYCLE 12 DAY 1; n=15, 13: number analyzed (Participants) | 15 | 13
  DBP; CYCLE 12 DAY 1; n=15, 13 | 0.6 (7.80) | 2.1 (8.65)
  DBP; CYCLE 13 DAY 1; n=13, 12: number analyzed (Participants) | 13 | 12
  DBP; CYCLE 13 DAY 1; n=13, 12 | -2.2 (6.07) | -2.7 (7.64)
  DBP; CYCLE 14 DAY 1; n=12, 12: number analyzed (Participants) | 12 | 12
  DBP; CYCLE 14 DAY 1; n=12, 12 | 0.7 (6.87) | 3.3 (11.78)
  DBP; CYCLE 15 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  DBP; CYCLE 15 DAY 1; n=10, 9 | 2.1 (8.49) | 1.1 (12.97)
  DBP; CYCLE 16 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  DBP; CYCLE 16 DAY 1; n=10, 9 | 0.1 (7.68) | 0.1 (11.88)
  DBP; CYCLE 17 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  DBP; CYCLE 17 DAY 1; n=8, 8 | -1.5 (8.23) | 5.0 (7.15)
  DBP; CYCLE 18 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  DBP; CYCLE 18 DAY 1; n=8, 8 | 0.1 (6.47) | 3.4 (11.15)
  DBP; CYCLE 19 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  DBP; CYCLE 19 DAY 1; n=6, 8 | -2.5 (5.82) | 5.5 (12.17)
  DBP; CYCLE 20 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  DBP; CYCLE 20 DAY 1; n=6, 8 | 2.3 (3.83) | 3.5 (10.09)
  DBP; CYCLE 21 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  DBP; CYCLE 21 DAY 1; n=4, 8 | 0.8 (2.99) | 2.8 (11.96)
  DBP; CYCLE 22 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  DBP; CYCLE 22 DAY 1; n=4, 8 | -1.8 (3.95) | 3.8 (7.63)
  DBP; CYCLE 23 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  DBP; CYCLE 23 DAY 1; n=4, 8 | 2.5 (4.20) | 5.1 (12.12)
  DBP; CYCLE 24 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  DBP; CYCLE 24 DAY 1; n=4, 8 | -3.0 (11.17) | 2.5 (12.99)
  DBP; CYCLE 25 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  DBP; CYCLE 25 DAY 1; n=4, 8 | 3.5 (3.11) | 2.5 (15.80)
  DBP; CYCLE 26 DAY 1; n=4, 7: number analyzed (Participants) | 4 | 7
  DBP; CYCLE 26 DAY 1; n=4, 7 | 0.0 (3.27) | 4.0 (14.57)
  DBP; CYCLE 27 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  DBP; CYCLE 27 DAY 1; n=4, 5 | -3.3 (4.72) | 3.6 (11.67)
  DBP; CYCLE 28 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  DBP; CYCLE 28 DAY 1; n=4, 5 | 2.0 (1.63) | 4.0 (14.21)
  DBP; CYCLE 29 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  DBP; CYCLE 29 DAY 1; n=3, 4 | 1.7 (10.41) | -2.0 (7.26)
  DBP; CYCLE 30 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  DBP; CYCLE 30 DAY 1; n=3, 4 | -0.3 (4.04) | -2.3 (6.60)
  DBP; CYCLE 31 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  DBP; CYCLE 31 DAY 1; n=3, 4 | 6.7 (7.64) | 0.5 (11.45)
  DBP; CYCLE 32 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  DBP; CYCLE 32 DAY 1; n=3, 4 | 2.7 (7.51) | -0.3 (7.76)
  DBP; CYCLE 33 DAY 1; n=2, 4: number analyzed (Participants) | 2 | 4
  DBP; CYCLE 33 DAY 1; n=2, 4 | 0.5 (7.78) | -2.5 (8.50)
  DBP; CYCLE 34 DAY 1; n=1, 4: number analyzed (Participants) | 1 | 4
  DBP; CYCLE 34 DAY 1; n=1, 4 | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point. | -1.8 (6.99)
  DBP; CYCLE 35 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  DBP; CYCLE 35 DAY 1; n=0, 4 |  | -3.0 (8.12)
  DBP; CYCLE 36 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  DBP; CYCLE 36 DAY 1; n=0, 4 |  | 1.5 (3.00)
  DBP; CYCLE 37 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  DBP; CYCLE 37 DAY 1; n=0, 3 |  | 1.7 (12.58)
  DBP; CYCLE 38 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  DBP; CYCLE 38 DAY 1; n=0, 3 |  | -2.3 (6.81)
  DBP; CYCLE 39 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  DBP; CYCLE 39 DAY 1; n=0, 3 |  | 0.3 (10.50)
  DBP; CYCLE 40 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 40 DAY 1; n=0, 2 |  | 0.0 (0.00)
  DBP; CYCLE 41 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 41 DAY 1; n=0, 2 |  | -7.5 (3.54)
  DBP; CYCLE 42 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 42 DAY 1; n=0, 2 |  | 0.0 (0.00)
  DBP; CYCLE 43 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 43 DAY 1; n=0, 2 |  | -7.5 (3.54)
  DBP; CYCLE 44 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 44 DAY 1; n=0, 2 |  | -2.5 (3.54)
  DBP; CYCLE 45 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 45 DAY 1; n=0, 2 |  | -7.5 (3.54)
  DBP; CYCLE 46 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 46 DAY 1; n=0, 2 |  | -5.0 (7.07)
  DBP; CYCLE 47 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 47 DAY 1; n=0, 2 |  | -3.0 (24.04)
  DBP; CYCLE 48 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 48 DAY 1; n=0, 2 |  | -5.0 (7.07)
  DBP; CYCLE 49 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 49 DAY 1; n=0, 2 |  | -12.5 (3.54)
  DBP; CYCLE 50 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 50 DAY 1; n=0, 2 |  | -5.0 (7.07)
  DBP; CYCLE 51 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 51 DAY 1; n=0, 2 |  | -5.0 (7.07)
  DBP; CYCLE 52 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 52 DAY 1; n=0, 2 |  | -10.0 (7.07)
  DBP; CYCLE 53 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 53 DAY 1; n=0, 2 |  | -7.5 (3.54)
  DBP; CYCLE 54 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  DBP; CYCLE 54 DAY 1; n=0, 2 |  | -5.0 (7.07)
  DBP; CYCLE 55 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 55 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 56 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 56 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 57 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 57 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 58 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 58 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 59 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 59 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 60 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 60 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 61 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 61 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 62 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 62 DAY 1; n=0, 1 |  | -13.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 63 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 63 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 64 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 64 DAY 1; n=0, 1 |  | -14.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 65 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 65 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 66 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 66 DAY 1; n=0, 1 |  | -17.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 67 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 67 DAY 1; n=0, 1 |  | -14.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 68 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 68 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 69 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 69 DAY 1; n=0, 1 |  | -17.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 70 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 70 DAY 1; n=0, 1 |  | -16.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 71 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 71 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 72 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 72 DAY 1; n=0, 1 |  | -19.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 73 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 73 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 74 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 74 DAY 1; n=0, 1 |  | -14.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  DBP; CYCLE 75 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  DBP; CYCLE 75 DAY 1; n=0, 1 |  | -17.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.

18. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was obtained on Day 1 of each cycle. Baseline is the last assessment prior to first dose. Change from Baseline is the value at indicated time point minus the value at Baseline. NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time point.
Time Frame: Baseline and Day 1 of Cycles 2 to 75 (each cycle of 21 days)
Population: As Treated Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Beats per minute
  Cycle 2 Day 1, n=46, 44: number analyzed (Participants) | 46 | 44
  Cycle 2 Day 1, n=46, 44 | 0.7 (8.32) | -1.8 (9.42)
  CYCLE 3 DAY 1, n=39, 35: number analyzed (Participants) | 39 | 35
  CYCLE 3 DAY 1, n=39, 35 | 1.7 (7.69) | -1.6 (6.78)
  CYCLE 4; DAY 1; n=33, 32: number analyzed (Participants) | 33 | 32
  CYCLE 4; DAY 1; n=33, 32 | 1.0 (10.09) | 1.9 (7.61)
  CYCLE 5 DAY 1; n=27, 26: number analyzed (Participants) | 27 | 26
  CYCLE 5 DAY 1; n=27, 26 | 1.3 (9.45) | 0.2 (10.65)
  CYCLE 6 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  CYCLE 6 DAY 1; n=24, 22 | 0.2 (10.37) | 0.3 (8.31)
  CYCLE 7 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  CYCLE 7 DAY 1; n=24, 22 | 2.0 (8.40) | -1.8 (8.80)
  CYCLE 8 DAY 1; n=22, 21: number analyzed (Participants) | 22 | 21
  CYCLE 8 DAY 1; n=22, 21 | 0.5 (7.70) | -0.4 (7.30)
  CYCLE 9 DAY 1; n=19, 16: number analyzed (Participants) | 19 | 16
  CYCLE 9 DAY 1; n=19, 16 | 2.1 (8.04) | 0.3 (7.10)
  CYCLE 10 DAY 1; n=18, 16: number analyzed (Participants) | 18 | 16
  CYCLE 10 DAY 1; n=18, 16 | 2.3 (8.62) | 0.5 (13.54)
  CYCLE 11 DAY 1; n=16, 15: number analyzed (Participants) | 16 | 15
  CYCLE 11 DAY 1; n=16, 15 | -0.8 (6.51) | -2.0 (9.88)
  CYCLE 12 DAY 1; n=15, 13: number analyzed (Participants) | 15 | 13
  CYCLE 12 DAY 1; n=15, 13 | -0.7 (4.28) | 0.2 (9.92)
  CYCLE 13 DAY 1; n=13, 12: number analyzed (Participants) | 13 | 12
  CYCLE 13 DAY 1; n=13, 12 | 0.9 (5.47) | 0.9 (9.77)
  CYCLE 14 DAY 1; n=12, 12: number analyzed (Participants) | 12 | 12
  CYCLE 14 DAY 1; n=12, 12 | 1.6 (7.03) | 3.1 (10.25)
  CYCLE 15 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  CYCLE 15 DAY 1; n=10, 9 | 5.6 (12.39) | 2.2 (8.51)
  CYCLE 16 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  CYCLE 16 DAY 1; n=10, 9 | 3.3 (7.06) | 0.7 (9.12)
  CYCLE 17 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  CYCLE 17 DAY 1; n=8, 8 | 3.1 (7.20) | 1.6 (10.23)
  CYCLE 18 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  CYCLE 18 DAY 1; n=8, 8 | 6.4 (8.68) | -0.5 (6.12)
  CYCLE 19 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  CYCLE 19 DAY 1; n=6, 8 | -2.5 (10.54) | 0.5 (9.78)
  CYCLE 20 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  CYCLE 20 DAY 1; n=6, 8 | 0.3 (6.38) | 0.9 (7.36)
  CYCLE 21 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 21 DAY 1; n=4, 8 | 0.5 (1.91) | -1.4 (10.28)
  CYCLE 22 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 22 DAY 1; n=4, 8 | 0.5 (1.91) | 3.0 (13.41)
  CYCLE 23 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 23 DAY 1; n=4, 8 | -3.8 (6.02) | 2.9 (9.76)
  CYCLE 24 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 24 DAY 1; n=4, 8 | -2.5 (5.97) | 2.9 (10.92)
  CYCLE 25 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 25 DAY 1; n=4, 8 | -1.8 (2.06) | 0.3 (11.13)
  CYCLE 26 DAY 1; n=4, 7: number analyzed (Participants) | 4 | 7
  CYCLE 26 DAY 1; n=4, 7 | -0.5 (1.91) | 1.6 (11.43)
  CYCLE 27 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  CYCLE 27 DAY 1; n=4, 5 | -2.0 (2.31) | 2.4 (11.70)
  CYCLE 28 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  CYCLE 28 DAY 1; n=4, 5 | -1.8 (5.56) | -0.2 (13.68)
  CYCLE 29 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 29 DAY 1; n=3, 4 | 0.0 (4.00) | -3.8 (6.45)
  CYCLE 30 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 30 DAY 1; n=3, 4 | 0.3 (2.08) | -9.3 (5.25)
  CYCLE 31 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 31 DAY 1; n=3, 4 | -2.7 (6.43) | -0.8 (8.77)
  CYCLE 32 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 32 DAY 1; n=3, 4 | 2.0 (4.00) | -3.8 (6.65)
  CYCLE 33 DAY 1; n=2, 4: number analyzed (Participants) | 2 | 4
  CYCLE 33 DAY 1; n=2, 4 | -2.0 (0.00) | -5.5 (7.55)
  CYCLE 34 DAY 1; n=1, 4: number analyzed (Participants) | 1 | 4
  CYCLE 34 DAY 1; n=1, 4 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point. | -3.5 (4.43)
  CYCLE 35 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  CYCLE 35 DAY 1; n=0, 4 |  | -4.8 (4.99)
  CYCLE 36 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  CYCLE 36 DAY 1; n=0, 4 |  | -8.0 (8.37)
  CYCLE 37 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 37 DAY 1; n=0, 3 |  | -9.3 (6.11)
  CYCLE 38 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 38 DAY 1; n=0, 3 |  | -2.0 (6.93)
  CYCLE 39 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 39 DAY 1; n=0, 3 |  | -4.7 (6.43)
  CYCLE 40 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 40 DAY 1; n=0, 2 |  | -4.0 (8.49)
  CYCLE 41 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 41 DAY 1; n=0, 2 |  | -7.0 (9.90)
  CYCLE 42 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 42 DAY 1; n=0, 2 |  | -2.0 (8.49)
  CYCLE 43 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 43 DAY 1; n=0, 2 |  | -6.0 (14.14)
  CYCLE 44 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 44 DAY 1; n=0, 2 |  | -2.0 (14.14)
  CYCLE 45 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 45 DAY 1; n=0, 2 |  | -4.0 (14.14)
  CYCLE 46 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 46 DAY 1; n=0, 2 |  | -3.0 (18.38)
  CYCLE 47 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 47 DAY 1; n=0, 2 |  | -2.0 (14.14)
  CYCLE 48 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 48 DAY 1; n=0, 2 |  | -3.0 (15.56)
  CYCLE 49 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 49 DAY 1; n=0, 2 |  | -9.0 (9.90)
  CYCLE 50 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 50 DAY 1; n=0, 2 |  | -5.0 (9.90)
  CYCLE 51 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 51 DAY 1; n=0, 2 |  | -5.0 (12.73)
  CYCLE 52 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 52 DAY 1; n=0, 2 |  | -8.0 (11.31)
  CYCLE 53 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 53 DAY 1; n=0, 2 |  | -10.0 (2.83)
  CYCLE 54 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 54 DAY 1; n=0, 2 |  | -2.0 (8.49)
  CYCLE 55 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 55 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 56 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 56 DAY 1; n=0, 1 |  | -12.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 57 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 57 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 58 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 58 DAY 1; n=0, 1 |  | -8.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 59 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 59 DAY 1; n=0, 1 |  | -12.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 60 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 60 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 61 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 61 DAY 1; n=0, 1 |  | -12.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 62 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 62 DAY 1; n=0, 1 |  | -14.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 63 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 63 DAY 1; n=0, 1 |  | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 64 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 64 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 65 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 65 DAY 1; n=0, 1 |  | -11.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 66 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 66 DAY 1; n=0, 1 |  | -12.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 67 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 67 DAY 1; n=0, 1 |  | -9.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 68 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 68 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 69 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 69 DAY 1; n=0, 1 |  | -12.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 70 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 70 DAY 1; n=0, 1 |  | -9.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 71 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 71 DAY 1; n=0, 1 |  | -7.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 72 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 72 DAY 1; n=0, 1 |  | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 73 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 73 DAY 1; n=0, 1 |  | -9.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 74 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 74 DAY 1; n=0, 1 |  | -8.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 75 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 75 DAY 1; n=0, 1 |  | -9.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.

19. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was obtained on Day 1 of each cycle. Baseline is the last assessment prior to first dose. Change from Baseline is the value at indicated time point minus the value at Baseline. NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time point.
Time Frame: Baseline and Day 1 of Cycles 2 to 75 (each cycle of 21 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Celsius
  Cycle 2 Day 1, n=46, 43: number analyzed (Participants) | 46 | 43
  Cycle 2 Day 1, n=46, 43 | 0.02 (0.288) | -0.02 (0.242)
  CYCLE 3 DAY 1, n=39, 35: number analyzed (Participants) | 39 | 35
  CYCLE 3 DAY 1, n=39, 35 | -0.01 (0.374) | -0.11 (0.340)
  CYCLE 4; DAY 1; n=33, 32: number analyzed (Participants) | 33 | 32
  CYCLE 4; DAY 1; n=33, 32 | 0.02 (0.354) | -0.05 (0.298)
  CYCLE 5 DAY 1; n=27, 26: number analyzed (Participants) | 27 | 26
  CYCLE 5 DAY 1; n=27, 26 | 0.05 (0.374) | -0.04 (0.218)
  CYCLE 6 DAY 1; n=23, 22: number analyzed (Participants) | 23 | 22
  CYCLE 6 DAY 1; n=23, 22 | -0.05 (0.374) | -0.07 (0.223)
  CYCLE 7 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  CYCLE 7 DAY 1; n=24, 22 | 0.03 (0.334) | -0.10 (0.408)
  CYCLE 8 DAY 1; n=21, 21: number analyzed (Participants) | 21 | 21
  CYCLE 8 DAY 1; n=21, 21 | 0.01 (0.460) | 0.02 (0.161)
  CYCLE 9 DAY 1; n=19, 16: number analyzed (Participants) | 19 | 16
  CYCLE 9 DAY 1; n=19, 16 | 0.04 (0.493) | 0.00 (0.171)
  CYCLE 10 DAY 1; n=18, 16: number analyzed (Participants) | 18 | 16
  CYCLE 10 DAY 1; n=18, 16 | 0.05 (0.539) | 0.04 (0.200)
  CYCLE 11 DAY 1; n=16, 15: number analyzed (Participants) | 16 | 15
  CYCLE 11 DAY 1; n=16, 15 | -0.02 (0.468) | -0.09 (0.181)
  CYCLE 12 DAY 1; n=15, 13: number analyzed (Participants) | 15 | 13
  CYCLE 12 DAY 1; n=15, 13 | 0.00 (0.270) | 0.02 (0.245)
  CYCLE 13 DAY 1; n=13, 12: number analyzed (Participants) | 13 | 12
  CYCLE 13 DAY 1; n=13, 12 | 0.00 (0.354) | 0.03 (0.176)
  CYCLE 14 DAY 1; n=12, 12: number analyzed (Participants) | 12 | 12
  CYCLE 14 DAY 1; n=12, 12 | 0.13 (0.380) | -0.04 (0.219)
  CYCLE 15 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  CYCLE 15 DAY 1; n=10, 9 | 0.11 (0.420) | -0.13 (0.269)
  CYCLE 16 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  CYCLE 16 DAY 1; n=10, 9 | 0.01 (0.318) | -0.04 (0.174)
  CYCLE 17 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  CYCLE 17 DAY 1; n=8, 8 | 0.00 (0.227) | 0.05 (0.076)
  CYCLE 18 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  CYCLE 18 DAY 1; n=8, 8 | -0.14 (0.346) | -0.09 (0.189)
  CYCLE 19 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  CYCLE 19 DAY 1; n=6, 8 | -0.10 (0.456) | 0.10 (0.207)
  CYCLE 20 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  CYCLE 20 DAY 1; n=6, 8 | -0.02 (0.397) | 0.01 (0.146)
  CYCLE 21 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 21 DAY 1; n=4, 8 | 0.13 (0.411) | -0.01 (0.304)
  CYCLE 22 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 22 DAY 1; n=4, 8 | 0.17 (0.206) | 0.00 (0.193)
  CYCLE 23 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 23 DAY 1; n=4, 8 | 0.03 (0.299) | 0.13 (0.231)
  CYCLE 24 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 24 DAY 1; n=4, 8 | 0.18 (0.171) | 0.06 (0.119)
  CYCLE 25 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 25 DAY 1; n=4, 8 | 0.20 (0.432) | 0.00 (0.185)
  CYCLE 26 DAY 1; n=4, 7: number analyzed (Participants) | 4 | 7
  CYCLE 26 DAY 1; n=4, 7 | 0.15 (0.129) | -0.01 (0.308)
  CYCLE 27 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  CYCLE 27 DAY 1; n=4, 5 | 0.18 (0.171) | 0.10 (0.173)
  CYCLE 28 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  CYCLE 28 DAY 1; n=4, 5 | 0.15 (0.208) | -0.02 (0.179)
  CYCLE 29 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 29 DAY 1; n=3, 4 | 0.13 (0.153) | -0.02 (0.275)
  CYCLE 30 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 30 DAY 1; n=3, 4 | 0.10 (0.173) | 0.00 (0.082)
  CYCLE 31 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 31 DAY 1; n=3, 4 | -0.07 (0.351) | 0.05 (0.265)
  CYCLE 32 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 32 DAY 1; n=3, 4 | 0.10 (0.173) | -0.05 (0.265)
  CYCLE 33 DAY 1; n=2, 4: number analyzed (Participants) | 2 | 4
  CYCLE 33 DAY 1; n=2, 4 | 0.30 (0.424) | -0.07 (0.222)
  CYCLE 34 DAY 1; n=1, 4: number analyzed (Participants) | 1 | 4
  CYCLE 34 DAY 1; n=1, 4 | 0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point | -0.20 (0.283)
  CYCLE 35 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  CYCLE 35 DAY 1; n=0, 4 |  | -0.05 (0.058)
  CYCLE 36 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  CYCLE 36 DAY 1; n=0, 4 |  | -0.07 (0.150)
  CYCLE 37 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 37 DAY 1; n=0, 3 |  | -0.30 (0.458)
  CYCLE 38 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 38 DAY 1; n=0, 3 |  | 0.00 (0.100)
  CYCLE 39 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 39 DAY 1; n=0, 3 |  | -0.07 (0.058)
  CYCLE 40 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 40 DAY 1; n=0, 2 |  | 0.00 (0.00)
  CYCLE 41 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 41 DAY 1; n=0, 2 |  | -0.10 (0.141)
  CYCLE 42 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 42 DAY 1; n=0, 2 |  | 0.05 (0.071)
  CYCLE 43 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 43 DAY 1; n=0, 2 |  | -0.05 (0.212)
  CYCLE 44 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 44 DAY 1; n=0, 2 |  | 0.00 (0.141)
  CYCLE 45 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 45 DAY 1; n=0, 2 |  | 0.00 (0.283)
  CYCLE 46 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 46 DAY 1; n=0, 2 |  | -0.05 (0.071)
  CYCLE 47 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 47 DAY 1; n=0, 2 |  | 0.05 (0.212)
  CYCLE 48 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 48 DAY 1; n=0, 2 |  | 0.00 (0.000)
  CYCLE 49 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 49 DAY 1; n=0, 2 |  | -0.05 (0.212)
  CYCLE 50 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 50 DAY 1; n=0, 2 |  | 0.00 (0.141)
  CYCLE 51 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 51 DAY 1; n=0, 2 |  | -0.05 (0.071)
  CYCLE 52 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 52 DAY 1; n=0, 2 |  | -0.10 (0.141)
  CYCLE 53 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 53 DAY 1; n=0, 2 |  | 0.05 (0.071)
  CYCLE 54 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 54 DAY 1; n=0, 2 |  | -0.05 (0.071)
  CYCLE 55 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 55 DAY 1; n=0, 1 |  | -0.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 56 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 56 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 57 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 57 DAY 1; n=0, 1 |  | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 58 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 58 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 59 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 59 DAY 1; n=0, 1 |  | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 60 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 60 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 61 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 61 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 62 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 62 DAY 1; n=0, 1 |  | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 63 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 63 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 64 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 64 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 65 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 65 DAY 1; n=0, 1 |  | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 66 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 66 DAY 1; n=0, 1 |  | -0.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 67 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 67 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 68 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 68 DAY 1; n=0, 1 |  | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 69 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 69 DAY 1; n=0, 1 |  | -0.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 70 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 70 DAY 1; n=0, 1 |  | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 71 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 71 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 72 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 72 DAY 1; n=0, 1 |  | -0.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 73 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 73 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 74 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 74 DAY 1; n=0, 1 |  | -0.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point
  CYCLE 75 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 75 DAY 1; n=0, 1 |  | -0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point

20. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was obtained on Day 1 of each cycle. Baseline is the last assessment prior to first dose.Change from Baseline is the value at indicated time point minus the value at Baseline. NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time point.
Time Frame: Baseline and Day 1 of Cycles 2 to 75 (each cycle of 21 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Breaths per minute
  CYCLE 2 Day 1, n=46, 44: number analyzed (Participants) | 46 | 44
  CYCLE 2 Day 1, n=46, 44 | -0.1 (1.62) | 0.1 (1.31)
  CYCLE 3 DAY 1, n=39, 35: number analyzed (Participants) | 39 | 35
  CYCLE 3 DAY 1, n=39, 35 | 0.2 (2.34) | -0.2 (1.71)
  CYCLE 4; DAY 1; n=32, 32: number analyzed (Participants) | 32 | 32
  CYCLE 4; DAY 1; n=32, 32 | 0.2 (1.79) | -0.3 (1.45)
  CYCLE 5 DAY 1; n=26, 26: number analyzed (Participants) | 26 | 26
  CYCLE 5 DAY 1; n=26, 26 | -0.1 (1.86) | -0.3 (1.50)
  CYCLE 6 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  CYCLE 6 DAY 1; n=24, 22 | 0.5 (2.15) | -0.3 (1.88)
  CYCLE 7 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  CYCLE 7 DAY 1; n=24, 22 | -0.1 (2.09) | -0.2 (1.74)
  CYCLE 8 DAY 1; n=21, 21: number analyzed (Participants) | 21 | 21
  CYCLE 8 DAY 1; n=21, 21 | 0.6 (1.78) | -0.1 (1.59)
  CYCLE 9 DAY 1; n=19, 16: number analyzed (Participants) | 19 | 16
  CYCLE 9 DAY 1; n=19, 16 | -0.5 (1.98) | -0.2 (2.04)
  CYCLE 10 DAY 1; n=18, 16: number analyzed (Participants) | 18 | 16
  CYCLE 10 DAY 1; n=18, 16 | -1.7 (2.95) | -0.4 (2.03)
  CYCLE 11 DAY 1; n=16, 15: number analyzed (Participants) | 16 | 15
  CYCLE 11 DAY 1; n=16, 15 | -0.8 (1.97) | -0.8 (2.21)
  CYCLE 12 DAY 1; n=15, 13: number analyzed (Participants) | 15 | 13
  CYCLE 12 DAY 1; n=15, 13 | 0.0 (2.48) | -1.0 (2.45)
  CYCLE 13 DAY 1; n=13, 12: number analyzed (Participants) | 13 | 12
  CYCLE 13 DAY 1; n=13, 12 | -0.2 (1.69) | -0.7 (2.67)
  CYCLE 14 DAY 1; n=12, 12: number analyzed (Participants) | 12 | 12
  CYCLE 14 DAY 1; n=12, 12 | 0.4 (2.43) | -1.0 (2.52)
  CYCLE 15 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  CYCLE 15 DAY 1; n=10, 9 | -0.5 (1.65) | -0.9 (3.06)
  CYCLE 16 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  CYCLE 16 DAY 1; n=10, 9 | -0.5 (1.72) | -0.9 (2.76)
  CYCLE 17 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  CYCLE 17 DAY 1; n=8, 8 | 0.0 (2.20) | 0.1 (1.81)
  CYCLE 18 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  CYCLE 18 DAY 1; n=8, 8 | -0.4 (2.07) | 0.4 (1.60)
  CYCLE 19 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  CYCLE 19 DAY 1; n=6, 8 | 0.7 (1.37) | 0.0 (1.51)
  CYCLE 20 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  CYCLE 20 DAY 1; n=6, 8 | 0.2 (0.75) | 0.0 (1.60)
  CYCLE 21 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 21 DAY 1; n=4, 8 | 0.8 (0.96) | -0.1 (1.64)
  CYCLE 22 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 22 DAY 1; n=4, 8 | 0.0 (0.00) | -0.1 (1.36)
  CYCLE 23 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 23 DAY 1; n=4, 8 | 0.5 (1.00) | 0.4 (1.60)
  CYCLE 24 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 24 DAY 1; n=4, 8 | -0.3 (1.26) | 0.0 (1.20)
  CYCLE 25 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 25 DAY 1; n=4, 8 | -0.3 (0.50) | -0.3 (1.49)
  CYCLE 26 DAY 1; n=4, 7: number analyzed (Participants) | 4 | 7
  CYCLE 26 DAY 1; n=4, 7 | -0.5 (1.00) | 0.0 (1.63)
  CYCLE 27 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  CYCLE 27 DAY 1; n=4, 5 | 0.0 (1.41) | 0.0 (1.00)
  CYCLE 28 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  CYCLE 28 DAY 1; n=4, 5 | -0.3 (0.50) | 0.2 (2.17)
  CYCLE 29 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 29 DAY 1; n=3, 4 | -0.7 (1.53) | -0.3 (2.22)
  CYCLE 30 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 30 DAY 1; n=3, 4 | 0.0 (0.00) | -0.3 (2.06)
  CYCLE 31 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 31 DAY 1; n=3, 4 | 0.7 (0.58) | 0.3 (2.36)
  CYCLE 32 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 32 DAY 1; n=3, 4 | -0.7 (1.53) | 0.0 (2.16)
  CYCLE 33 DAY 1; n=2, 4: number analyzed (Participants) | 2 | 4
  CYCLE 33 DAY 1; n=2, 4 | -2.0 (0.00) | -0.8 (1.50)
  CYCLE 34 DAY 1; n=1, 4: number analyzed (Participants) | 1 | 4
  CYCLE 34 DAY 1; n=1, 4 | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point. | 0.8 (1.50)
  CYCLE 35 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  CYCLE 35 DAY 1; n=0, 4 |  | 0.0 (1.83)
  CYCLE 36 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  CYCLE 36 DAY 1; n=0, 4 |  | 0.3 (1.71)
  CYCLE 37 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 37 DAY 1; n=0, 3 |  | -1.0 (1.73)
  CYCLE 38 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 38 DAY 1; n=0, 3 |  | -0.3 (2.52)
  CYCLE 39 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 39 DAY 1; n=0, 3 |  | -1.0 (1.73)
  CYCLE 40 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 40 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 41 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 41 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 42 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 42 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 43 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 43 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 44 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 44 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 45 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 45 DAY 1; n=0, 2 |  | -1.5 (0.71)
  CYCLE 46 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 46 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 47 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 47 DAY 1; n=0, 2 |  | -0.5 (0.71)
  CYCLE 48 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 48 DAY 1; n=0, 2 |  | 1.0 (1.41)
  CYCLE 49 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 49 DAY 1; n=0, 2 |  | -1.0 (1.41)
  CYCLE 50 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 50 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 51 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 51 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 52 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 52 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 53 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 53 DAY 1; n=0, 2 |  | -1.0 (1.41)
  CYCLE 54 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 54 DAY 1; n=0, 2 |  | 0.0 (0.00)
  CYCLE 55 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 55 DAY 1; n=0, 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 56 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 56 DAY 1; n=0, 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 57 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 57 DAY 1; n=0, 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 58 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 58 DAY 1; n=0, 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 59 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 59 DAY 1; n=0, 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 60 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 60 DAY 1; n=0, 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 61 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 61 DAY 1; n=0, 1 |  | 0.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 62 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 62 DAY 1; n=0, 1 |  | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 63 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 63 DAY 1; n=0, 1 |  | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 64 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 64 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 65 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 65 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 66 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 66 DAY 1; n=0, 1 |  | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 67 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 67 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 68 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 68 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 69 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 69 DAY 1; n=0, 1 |  | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 70 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 70 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 71 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 71 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 72 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 72 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 73 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 73 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 74 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 74 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 75 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 75 DAY 1; n=0, 1 |  | -2.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.

21. Secondary Outcome: Change From Baseline in Weight
Description: Weight was obtained on Day 1 of each cycle. Baseline is the last assessment prior to first dose. Change from Baseline is the value at indicated time point minus the value at Baseline. NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time point.
Time Frame: Baseline and Day 1 of Cycles 2 to 75 (each cycle of 21 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 51 | 50
Kilograms
  Cycle 2 Day 1, n=46, 44: number analyzed (Participants) | 46 | 44
  Cycle 2 Day 1, n=46, 44 | -1.51 (2.192) | -1.55 (2.405)
  CYCLE 3 DAY 1, n=39, 35: number analyzed (Participants) | 39 | 35
  CYCLE 3 DAY 1, n=39, 35 | -2.54 (2.734) | -1.88 (2.710)
  CYCLE 4; DAY 1; n=33, 32: number analyzed (Participants) | 33 | 32
  CYCLE 4; DAY 1; n=33, 32 | -3.02 (2.451) | -1.86 (3.305)
  CYCLE 5 DAY 1; n=27, 26: number analyzed (Participants) | 27 | 26
  CYCLE 5 DAY 1; n=27, 26 | -3.31 (2.521) | -2.01 (3.301)
  CYCLE 6 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  CYCLE 6 DAY 1; n=24, 22 | -3.25 (3.078) | -2.61 (4.200)
  CYCLE 7 DAY 1; n=24, 22: number analyzed (Participants) | 24 | 22
  CYCLE 7 DAY 1; n=24, 22 | -3.75 (4.172) | -2.14 (5.877)
  CYCLE 8 DAY 1; n=22, 21: number analyzed (Participants) | 22 | 21
  CYCLE 8 DAY 1; n=22, 21 | -3.89 (4.384) | -2.61 (5.016)
  CYCLE 9 DAY 1; n=19, 16: number analyzed (Participants) | 19 | 16
  CYCLE 9 DAY 1; n=19, 16 | -4.14 (5.151) | -2.14 (4.998)
  CYCLE 10 DAY 1; n=18, 16: number analyzed (Participants) | 18 | 16
  CYCLE 10 DAY 1; n=18, 16 | -5.50 (6.983) | -1.99 (5.478)
  CYCLE 11 DAY 1; n=16, 15: number analyzed (Participants) | 16 | 15
  CYCLE 11 DAY 1; n=16, 15 | -5.70 (6.045) | -1.67 (4.681)
  CYCLE 12 DAY 1; n=15, 13: number analyzed (Participants) | 15 | 13
  CYCLE 12 DAY 1; n=15, 13 | -5.85 (5.206) | -1.72 (4.260)
  CYCLE 13 DAY 1; n=13, 12: number analyzed (Participants) | 13 | 12
  CYCLE 13 DAY 1; n=13, 12 | -6.54 (5.795) | -1.11 (4.483)
  CYCLE 14 DAY 1; n=12, 12: number analyzed (Participants) | 12 | 12
  CYCLE 14 DAY 1; n=12, 12 | -7.03 (6.500) | -1.23 (3.899)
  CYCLE 15 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  CYCLE 15 DAY 1; n=10, 9 | -7.21 (7.449) | -1.09 (4.705)
  CYCLE 16 DAY 1; n=10, 9: number analyzed (Participants) | 10 | 9
  CYCLE 16 DAY 1; n=10, 9 | -7.59 (6.970) | -0.93 (4.519)
  CYCLE 17 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  CYCLE 17 DAY 1; n=8, 8 | -8.49 (8.606) | -1.24 (5.205)
  CYCLE 18 DAY 1; n=8, 8: number analyzed (Participants) | 8 | 8
  CYCLE 18 DAY 1; n=8, 8 | -8.25 (9.002) | -0.80 (4.888)
  CYCLE 19 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  CYCLE 19 DAY 1; n=6, 8 | -8.78 (9.953) | -0.19 (5.044)
  CYCLE 20 DAY 1; n=6, 8: number analyzed (Participants) | 6 | 8
  CYCLE 20 DAY 1; n=6, 8 | -9.22 (10.752) | -0.40 (5.986)
  CYCLE 21 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 21 DAY 1; n=4, 8 | -3.03 (7.950) | -0.29 (6.354)
  CYCLE 22 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 22 DAY 1; n=4, 8 | -3.50 (7.735) | -0.32 (5.370)
  CYCLE 23 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 23 DAY 1; n=4, 8 | -4.13 (8.189) | -0.16 (5.297)
  CYCLE 24 DAY 1; n=4, 7: number analyzed (Participants) | 4 | 7
  CYCLE 24 DAY 1; n=4, 7 | -3.38 (7.273) | -1.93 (1.511)
  CYCLE 25 DAY 1; n=4, 8: number analyzed (Participants) | 4 | 8
  CYCLE 25 DAY 1; n=4, 8 | -3.88 (8.250) | 0.04 (5.789)
  CYCLE 26 DAY 1; n=4, 7: number analyzed (Participants) | 4 | 7
  CYCLE 26 DAY 1; n=4, 7 | -3.88 (6.981) | 0.54 (6.484)
  CYCLE 27 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  CYCLE 27 DAY 1; n=4, 5 | -4.88 (6.408) | -2.04 (2.308)
  CYCLE 28 DAY 1; n=4, 5: number analyzed (Participants) | 4 | 5
  CYCLE 28 DAY 1; n=4, 5 | -5.13 (6.115) | -2.20 (1.989)
  CYCLE 29 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 29 DAY 1; n=3, 4 | -5.50 (7.697) | -2.18 (1.786)
  CYCLE 30 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 30 DAY 1; n=3, 4 | -5.83 (7.286) | -3.25 (0.379)
  CYCLE 31 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 31 DAY 1; n=3, 4 | -5.50 (7.467) | -3.38 (0.435)
  CYCLE 32 DAY 1; n=3, 4: number analyzed (Participants) | 3 | 4
  CYCLE 32 DAY 1; n=3, 4 | -5.50 (7.467) | -3.05 (0.100)
  CYCLE 33 DAY 1; n=2, 4: number analyzed (Participants) | 2 | 4
  CYCLE 33 DAY 1; n=2, 4 | -1.75 (1.061) | -3.13 (0.150)
  CYCLE 34 DAY 1; n=1, 4: number analyzed (Participants) | 1 | 4
  CYCLE 34 DAY 1; n=1, 4 | -2.50 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point. | -3.18 (0.350)
  CYCLE 35 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  CYCLE 35 DAY 1; n=0, 4 |  | -3.25 (0.379)
  CYCLE 36 DAY 1; n=0, 4: number analyzed (Participants) | 0 | 4
  CYCLE 36 DAY 1; n=0, 4 |  | -3.38 (0.624)
  CYCLE 37 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 37 DAY 1; n=0, 3 |  | -3.17 (0.961)
  CYCLE 38 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 38 DAY 1; n=0, 3 |  | -2.63 (0.814)
  CYCLE 39 DAY 1; n=0, 3: number analyzed (Participants) | 0 | 3
  CYCLE 39 DAY 1; n=0, 3 |  | -3.00 (0.200)
  CYCLE 40 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 40 DAY 1; n=0, 2 |  | -3.40 (0.566)
  CYCLE 41 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 41 DAY 1; n=0, 2 |  | -2.90 (0.141)
  CYCLE 42 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 42 DAY 1; n=0, 2 |  | -3.00 (0.000)
  CYCLE 43 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 43 DAY 1; n=0, 2 |  | -2.90 (0.141)
  CYCLE 44 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 44 DAY 1; n=0, 2 |  | -3.90 (1.273)
  CYCLE 45 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 45 DAY 1; n=0, 2 |  | -4.40 (1.980)
  CYCLE 46 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 46 DAY 1; n=0, 2 |  | -3.90 (1.273)
  CYCLE 47 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 47 DAY 1; n=0, 2 |  | -3.40 (0.566)
  CYCLE 48 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 48 DAY 1; n=0, 2 |  | -3.65 (0.919)
  CYCLE 49 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 49 DAY 1; n=0, 2 |  | -4.40 (1.980)
  CYCLE 50 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 50 DAY 1; n=0, 2 |  | -4.15 (1.626)
  CYCLE 51 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 51 DAY 1; n=0, 2 |  | -3.65 (0.919)
  CYCLE 52 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 52 DAY 1; n=0, 2 |  | -2.90 (0.141)
  CYCLE 53 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 53 DAY 1; n=0, 2 |  | -4.40 (1.980)
  CYCLE 54 DAY 1; n=0, 2: number analyzed (Participants) | 0 | 2
  CYCLE 54 DAY 1; n=0, 2 |  | -3.65 (0.919)
  CYCLE 55 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 55 DAY 1; n=0, 1 |  | -2.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 56 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 56 DAY 1; n=0, 1 |  | -1.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 57 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 57 DAY 1; n=0, 1 |  | -0.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 58 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 58 DAY 1; n=0, 1 |  | -1.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 59 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 59 DAY 1; n=0, 1 |  | -0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 60 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 60 DAY 1; n=0, 1 |  | -0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 61 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 61 DAY 1; n=0, 1 |  | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 62 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 62 DAY 1; n=0, 1 |  | -0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 63 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 63 DAY 1; n=0, 1 |  | -0.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 64 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 64 DAY 1; n=0, 1 |  | -0.60 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 65 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 65 DAY 1; n=0, 1 |  | -2.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 66 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 66 DAY 1; n=0, 1 |  | -3.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 67 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 67 DAY 1; n=0, 1 |  | -3.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 68 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 68 DAY 1; n=0, 1 |  | -1.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 69 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 69 DAY 1; n=0, 1 |  | -1.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 70 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 70 DAY 1; n=0, 1 |  | 0.20 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 71 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 71 DAY 1; n=0, 1 |  | -0.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 72 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 72 DAY 1; n=0, 1 |  | -0.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 73 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 73 DAY 1; n=0, 1 |  | -1.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 74 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 74 DAY 1; n=0, 1 |  | -0.80 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 75 DAY 1; n=0, 1: number analyzed (Participants) | 0 | 1
  CYCLE 75 DAY 1; n=0, 1 |  | -0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.

22. Secondary Outcome: Serum Concentration of Mapatumumab
Description: Blood samples were collected for determination of serum mapatumumab concentration at the indicated time points. NA indicates standard deviation could not be calculated as only one participant was analyzed at the specified time points.
Time Frame: Day1 pre-dose(Cycle 1,2,4,5,6,8,9,10,12,14,16,17,18,20,22,24,26,28,30,32,34);end of infusion (Cycle 1);Day8 pre-dose(Cycle 1);Day15 pre-dose (Cycle 1,2);Day21(Cycle 2,4,6,8,9,12,14,16,18,20,22,24,26,28,30,32,34);Cycle 99(end of treatment) (21-day cycles)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Sorafenib+Mapatumumab 30 mg/kg
Number analyzed (Participants) | 50
Nanograms per milliliter
  CYCLE 1 Day 1, pre-dose, n=46: number analyzed (Participants) | 46
  CYCLE 1 Day 1, pre-dose, n=46 | 638.4 (2668.01)
  CYCLE 1 DAY 1,end of infusion, n=46: number analyzed (Participants) | 46
  CYCLE 1 DAY 1,end of infusion, n=46 | 555157.6 (260848.85)
  CYCLE 1; DAY 8, pre-dose; n=40: number analyzed (Participants) | 40
  CYCLE 1; DAY 8, pre-dose; n=40 | 250229.9 (89714.76)
  CYCLE 1 DAY 15, pre-dose; n=1: number analyzed (Participants) | 1
  CYCLE 1 DAY 15, pre-dose; n=1 | 121556.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 2 DAY 1, pre-dose; n=40: number analyzed (Participants) | 40
  CYCLE 2 DAY 1, pre-dose; n=40 | 126588.4 (149231.45)
  CYCLE 2 DAY 15, pre-dose; n=3: number analyzed (Participants) | 3
  CYCLE 2 DAY 15, pre-dose; n=3 | 128839.0 (153667.78)
  CYCLE 2 DAY 21; n=28: number analyzed (Participants) | 28
  CYCLE 2 DAY 21; n=28 | 180606.6 (109893.28)
  CYCLE 4 DAY 1, pre-dose; n=31: number analyzed (Participants) | 31
  CYCLE 4 DAY 1, pre-dose; n=31 | 194936.8 (142242.80)
  CYCLE 4, DAY 21; n=23: number analyzed (Participants) | 23
  CYCLE 4, DAY 21; n=23 | 183754.3 (93584.71)
  CYCLE 5, DAY 1, pre-dose; n=1: number analyzed (Participants) | 1
  CYCLE 5, DAY 1, pre-dose; n=1 | 223681.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 6, DAY 1, pre-dose; n=21: number analyzed (Participants) | 21
  CYCLE 6, DAY 1, pre-dose; n=21 | 160741.5 (64893.03)
  CYCLE 6, DAY 21; n=20: number analyzed (Participants) | 20
  CYCLE 6, DAY 21; n=20 | 201237.7 (75352.54)
  CYCLE 8, DAY 1, pre-dose; n=21: number analyzed (Participants) | 21
  CYCLE 8, DAY 1, pre-dose; n=21 | 246616.5 (204363.04)
  CYCLE 8, DAY 21; n=17: number analyzed (Participants) | 17
  CYCLE 8, DAY 21; n=17 | 187927.6 (104803.16)
  CYCLE 9, DAY 1, pre-dose; n=1: number analyzed (Participants) | 1
  CYCLE 9, DAY 1, pre-dose; n=1 | 136122.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 10, DAY 1, pre-dose; n=16: number analyzed (Participants) | 16
  CYCLE 10, DAY 1, pre-dose; n=16 | 204147.1 (103243.21)
  CYCLE 10, DAY 21; n=15: number analyzed (Participants) | 15
  CYCLE 10, DAY 21; n=15 | 219503.0 (105968.15)
  CYCLE 12, DAY 1, pre-dose; n=12: number analyzed (Participants) | 12
  CYCLE 12, DAY 1, pre-dose; n=12 | 200141.1 (93093.68)
  CYCLE 12, DAY 21; n=11: number analyzed (Participants) | 11
  CYCLE 12, DAY 21; n=11 | 256924.5 (111904.82)
  CYCLE 14, DAY 1, pre-dose; n=9: number analyzed (Participants) | 9
  CYCLE 14, DAY 1, pre-dose; n=9 | 207930.6 (84247.04)
  CYCLE 14, DAY 21 n=9: number analyzed (Participants) | 9
  CYCLE 14, DAY 21 n=9 | 256779.4 (127463.67)
  CYCLE 16, DAY 1, pre-dose; n=9: number analyzed (Participants) | 9
  CYCLE 16, DAY 1, pre-dose; n=9 | 196074.3 (100377.45)
  CYCLE 16, DAY 21; n=8: number analyzed (Participants) | 8
  CYCLE 16, DAY 21; n=8 | 253521.0 (87675.77)
  CYCLE 17, DAY 1, pre-dose; n=1: number analyzed (Participants) | 1
  CYCLE 17, DAY 1, pre-dose; n=1 | 156161.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 18, DAY 1, pre-dose; n=8: number analyzed (Participants) | 8
  CYCLE 18, DAY 1, pre-dose; n=8 | 199379.4 (61011.54)
  CYCLE 18, DAY 21; n=7: number analyzed (Participants) | 7
  CYCLE 18, DAY 21; n=7 | 229539.1 (86440.46)
  CYCLE 20 DAY 1, pre-dose; n=8: number analyzed (Participants) | 8
  CYCLE 20 DAY 1, pre-dose; n=8 | 189486.6 (54097.82)
  CYCLE 20, DAY 21; n=7: number analyzed (Participants) | 7
  CYCLE 20, DAY 21; n=7 | 222443.7 (86046.38)
  CYCLE 22 DAY 1, pre-dose; n=8: number analyzed (Participants) | 8
  CYCLE 22 DAY 1, pre-dose; n=8 | 208485.4 (80252.29)
  CYCLE 22, DAY 21; n=7: number analyzed (Participants) | 7
  CYCLE 22, DAY 21; n=7 | 212481.1 (110103.79)
  CYCLE 24 DAY 1, pre-dose; n=8: number analyzed (Participants) | 8
  CYCLE 24 DAY 1, pre-dose; n=8 | 219439.8 (71740.01)
  CYCLE 24, DAY 21; n=7: number analyzed (Participants) | 7
  CYCLE 24, DAY 21; n=7 | 221249.1 (73317.41)
  CYCLE 26 DAY 1, pre-dose; n=4: number analyzed (Participants) | 4
  CYCLE 26 DAY 1, pre-dose; n=4 | 223427.3 (67101.56)
  CYCLE 26, DAY 21; n=4: number analyzed (Participants) | 4
  CYCLE 26, DAY 21; n=4 | 295941.5 (100208.45)
  CYCLE 28 DAY 1, pre-dose; n=3: number analyzed (Participants) | 3
  CYCLE 28 DAY 1, pre-dose; n=3 | 219802.7 (115484.98)
  CYCLE 28, DAY 21; n=2: number analyzed (Participants) | 2
  CYCLE 28, DAY 21; n=2 | 173018.5 (54870.78)
  CYCLE 30 DAY 1, pre-dose; n=2: number analyzed (Participants) | 2
  CYCLE 30 DAY 1, pre-dose; n=2 | 173200.5 (13447.05)
  CYCLE 30, DAY 21; n=2: number analyzed (Participants) | 2
  CYCLE 30, DAY 21; n=2 | 180484.5 (14783.48)
  CYCLE 32 DAY 1, pre-dose; n=1: number analyzed (Participants) | 1
  CYCLE 32 DAY 1, pre-dose; n=1 | 178275.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 32, DAY 21; n=1: number analyzed (Participants) | 1
  CYCLE 32, DAY 21; n=1 | 177496.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 34 DAY 1, pre-dose; n=1: number analyzed (Participants) | 1
  CYCLE 34 DAY 1, pre-dose; n=1 | 150553.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 34, DAY 21; n=1: number analyzed (Participants) | 1
  CYCLE 34, DAY 21; n=1 | 134781.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed at the specified time point.
  CYCLE 99, end of treatment; n=14: number analyzed (Participants) | 14
  CYCLE 99, end of treatment; n=14 | 86640.1 (64981.14)

ADVERSE EVENTS:
Time Frame: Start of study treatment up to maximum of 52.9 months
Description: Treatment-emergent non-serious AEs and SAEs were collected in the As-Treated Population which comprised of participants who received at least part of 1 dose of study agent analyzed according to the treatment that they actually received.
Arm/Group | Sorafenib+Placebo | Sorafenib+Mapatumumab 30 mg/kg
All-Cause Mortality (participants affected / at risk) | 40/51 | 39/50
Serious Adverse Events (participants affected / at risk) | 27/51 | 21/50
Other Adverse Events (participants affected / at risk) | 47/51 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib+Placebo (N=51) | Sorafenib+Mapatumumab 30 mg/kg (N=50)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 3 (4)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 4 (4)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib+Placebo (N=51) | Sorafenib+Mapatumumab 30 mg/kg (N=50)
Anaemia (Blood and lymphatic system disorders) | 10 (15) | 8 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (9) | 7 (13)
Diarrhoea (Gastrointestinal disorders) | 19 (46) | 16 (29)
Abdominal pain (Gastrointestinal disorders) | 9 (22) | 8 (11)
Nausea (Gastrointestinal disorders) | 8 (11) | 8 (10)
Vomiting (Gastrointestinal disorders) | 7 (23) | 5 (7)
Ascites (Gastrointestinal disorders) | 6 (11) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (5)
Haemorrhoids (Gastrointestinal disorders) | 4 (5) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (4) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 15 (24) | 6 (10)
Asthenia (General disorders) | 8 (12) | 11 (26)
Oedema peripheral (General disorders) | 9 (12) | 6 (7)
Pyrexia (General disorders) | 3 (3) | 5 (8)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3) | 5 (7)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 3 (6)
Jaundice hepatocellular (Hepatobiliary disorders) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 22 (41) | 19 (34)
Lipase increased (Investigations) | 12 (37) | 17 (46)
Aspartate aminotransferase increased (Investigations) | 11 (37) | 9 (25)
Gamma-glutamyltransferase increased (Investigations) | 11 (17) | 8 (12)
Blood bilirubin increased (Investigations) | 9 (36) | 5 (14)
Alanine aminotransferase increased (Investigations) | 8 (18) | 7 (11)
Amylase increased (Investigations) | 8 (12) | 7 (29)
Platelet count decreased (Investigations) | 6 (34) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 5 (11) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 3 (3)
Weight increased (Investigations) | 0 (0) | 3 (4)
White blood cell count decreased (Investigations) | 3 (34) | 3 (9)
Decreased appetite (Metabolism and nutrition disorders) | 12 (17) | 9 (15)
Hypocalcaemia (Metabolism and nutrition disorders) | 9 (32) | 4 (15)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (9) | 7 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (20) | 3 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (7) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 4 (5) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 18 (29) | 19 (28)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (13)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (6)
Hypertension (Vascular disorders) | 12 (16) | 16 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT01258608/Prot_000.pdf
  • Statistical Analysis Plan (2011-11-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT01258608/SAP_001.pdf